CLINICAL TRIAL: NCT03102073
Title: Validation of Romanian Version of Radner Reading Charts
Status: Completed | Type: Observational
Sponsor: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Other Study IDs: OPRAD/0116/MD
Record Dates: First submitted 2017-03-17; First posted 2017-04-05 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-03

CONDITIONS: Visual Acuity
Keywords: Reading speed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radner test: reading speed evaluation
  Interventions: Diagnostic Test: Radner test

INTERVENTIONS:
Diagnostic Test: Radner test — * The A5 reading booklet is held by the subject
  * The subject is instructed to read sentence by sentence, by turning consecutively the pages of the booklet (on the first side is the number of sentence and the backward side contains the sentence)
  * The subject is instructed to read the sentences aloud as quickly and accurately as possible to the end, and to not correct reading errors.
  * One assessor is writing the reading time and records any reading errors on the scoring sheet while the second assessor is audio recording the operation
  * Stop criterion: reading time longer than 20 seconds or severe errors.
  Other Names: Validation of the Romanian version-Radner Reading Charts

SUMMARY:
Interventional, parallel groups, single center trial with a prospective design

DETAILED DESCRIPTION:
The "Radner Reading Charts" have been developed on the basis of the concept of "sentence optotypes" for the standardized examination of reading acuity and reading speed. Print sizes are logarithmically scaled (LogRAD) to permit statistical analysis, and the results obtained can be compared to other logarithmically scaled vision systems (e.g., LogMAR). To guarantee accurate, reproducible and standardized measurements of reading acuity and reading speed at every viewing distance, "sentence optotypes" have been created to minimize the variations between the test items and to keep the geometric proportions as constant as possible at all distances. Through interdisciplinary cooperation, a series of test sentences were developed that are highly comparable in terms of the number of words (14 words), as well as the word length, number of syllables, position of words, lexical difficulty and syntactical complexity. The most similar sentences were statistically selected for the Radner Reading Charts.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥18 years
* Visual acuity ≥ 20/20 Snellen in each eye
* Average daily reading time for students 5-7 hours and for non-students 0,5-2 hours
* Willingness to provide signed informed consent

Exclusion Criteria:

* Ocular pathologies that can influence the study results
* Alcohol ingestion
* Concomitant medication that can influence visual acuity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Reading speed | 2-4 months postsurgery
  in words per minute

SECONDARY OUTCOMES:
Reading errors | 2-4 months postsurgery
  count errors at each sentence

CONTACTS AND LOCATIONS:
Overall Officials: Serban Rosu, MD, Study Director — OPERA CRO
Locations (1):
- Opera Contract Research Organization Srl, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No